CLINICAL TRIAL: NCT01361555
Title: A Multicenter, Double-Blind, 58 Week Rollover Study to Assess the Safety and Tolerability of BMS-820836 in Patients With Treatment Resistant Major Depression
Brief Title: Long-term Safety and Tolerability of BMS-820836 in the Treatment of Patients With Treatment Resistant Major Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to meet primary endpoint
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN162-010; 2010-024371-12 (EudraCT Number)
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Placebo + BMS-820836 (0.5 mg/day) (Experimental)
  Interventions: Drug: Placebo matching with BMS-820836; Drug: BMS-820836
- Arm 2: Placebo + BMS-820836 (1 mg/day) (Experimental)
  Interventions: Drug: Placebo matching with BMS-820836; Drug: BMS-820836
- Arm 3: Placebo + BMS-820836 (2 mg/day) (Experimental)
  Interventions: Drug: Placebo matching with BMS-820836; Drug: BMS-820836

INTERVENTIONS:
Drug: Placebo matching with BMS-820836 — Tablet, Oral, 0.0 mg, Once daily, 54 weeks
Drug: BMS-820836 — Tablet, Oral, 0.5 mg, Once daily, 54 weeks
  Arms: Arm 1: Placebo + BMS-820836 (0.5 mg/day)
Drug: BMS-820836 — Tablet, Oral, 1.0 mg, Once daily, 54 weeks
  Arms: Arm 2: Placebo + BMS-820836 (1 mg/day)
Drug: BMS-820836 — Tablet, Oral, 2.0 mg, Once daily, 54 weeks
  Arms: Arm 3: Placebo + BMS-820836 (2 mg/day)

SUMMARY:
The purpose of this study it to evaluate the long-term safety and tolerability of BMS-820836 in patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of age 18-65 years (Argentina the minimum age will be 24 years of age)
* Patients randomized in parent study who complete CN162-006 and CN162-007 who consent to enter the rollover study.
* Patient not randomized in parent study that meet inadequate response criteria

Exclusion Criteria:

* Patients who represent a significant risk of committing suicide based on the clinical judgment of the investigator, history or routine psychiatric status exam.
* Patients with a Cardiovascular System Organ Class adverse event(s) occurring in parent study (CN162-006 or CN162-007), that in the investigators judgment is clinically significant and would impact safety of the subject in the current study [including but not limited to left bundle branch block, or prolonged QT interval corrected (QTc)].
* In addition, patients should be excluded if they have any laboratory test, vital sign, electrocardiogram (ECG) or clinical findings that in the investigator's judgment is clinically significantly abnormal and could impact the safety of the patient or the interpretation of study assessments in the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Long-term effects of BMS-820836 on blood pressure in patients with depression | Baseline through Week 54

SECONDARY OUTCOMES:
• Adverse Events (AEs), Serious Adverse Events, and Discontinuations Due to AEs | Baseline through Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (136):
- United States (93):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - K & S Professional Research Services, Llc, Little Rock, Arkansas
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Catalina Research Institute, Llc, Chino, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Behavioral Research Specialists, Llc, Glendale, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Neuropsychiatric Research Center Of Orange County, Orange, California
  - Pacific Clinical Research Medical Group, Orange, California
  - Anderson Clinical Research, Redlands, California
  - California Neuropsychopharmacology Clinical, San Diego, California
  - Pacific Research Network, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - Artemis Institute For Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Meridien Research, Brooksville, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Amit Vijapura, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, Llc, Orlando, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Institute Of Medicine & Research, Atlanta, Georgia
  - Comprehensive Clinical Development, Inc, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Alpine Clinic, Lafayette, Indiana
  - Clinco, Terre Haute, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - James G. Barbee, Md, Llc, New Orleans, Louisiana
  - J. Gary Booker, Md, Apmc, Shreveport, Louisiana
  - Mclean Hospital, Belmont, Massachusetts
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Spri Clinical Trials, Llc, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Comprehensive Clinical Development, Inc, Jamaica, New York
  - Village Clinical Research, Inc., New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Richard H. Weisler, Md, Pa & Assoc., Raleigh, North Carolina
  - Northcoast Clinical Trials, Inc, Beachwood, Ohio
  - Patient Priority Clinical Sites, Llc, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology & Neuroscience Center Of Ohio, Toledo, Ohio
  - Ips Research Company, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Oregon Center For Clinical Investigations, Inc. (Occi, Inc), Portland, Oregon
  - Summit Research Network (Oregon) Inc, Portland, Oregon
  - Oregon Center For Clinical Investigations, Inc (Occi, Inc), Salem, Oregon
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, Llc, Norristown, Pennsylvania
  - Univ Of Penn, Philadelphia, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Comprehensive Psychiatric Care, Pittsburgh, Pennsylvania
  - Bioscience Research, Llc, Pittsburgh, Pennsylvania
  - Insite Clinical Research, Pittsburgh, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Research Services, Columbia, South Carolina
  - Psychiatric Consultants, Pc, Franklin, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Futuresearch Trials, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - Futuresearch Trials Of Dallas, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Ut Health-Houston, Houston, Texas
  - Red Oak Psychiatry Associates, Pa, Houston, Texas
  - San Antonio Psychiatric Research Center, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Ericksen Research And Development, Clinton, Utah
  - Radiant Research, Inc., Murray, Utah
  - Psychiatric And Behavioral Solutions, Salt Lake City, Utah
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) Llc, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin
  - Independent Psychiatric Consultants, Sc, Dba, Ipc Research, Waukesha, Wisconsin
- Argentina (4):
  - Local Institution, Caba, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Mendoza, Mendoza Province
- Australia (4):
  - Local Institution, Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Nedlands, Western Australia
- Local Institution, Vienna, Austria
- Finland (6):
  - Local Institution, Helsinki
  - Local Institution, Jarvenpaa
  - Local Institution, Oulu
  - Local Institution, Seinäjoki
  - Local Institution, Tampere
  - Local Institution, Turku
- France (7):
  - Local Institution, Montpellier, France
  - Local Institution, Paris, France
  - Local Institution, Dole
  - Local Institution, Douai
  - Local Institution, Élancourt
  - Local Institution, Jonzac
  - Local Institution, Limoges
- India (7):
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Chennai
  - Local Institution, Pune
  - Local Institution, Varanasi
  - Local Institution, Vishakapattanam
- Italy (2):
  - Local Institution, Pisa
  - Local Institution, Siena
- Local Institution, Ponce, Puerto Rico
- South Africa (4):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
- Spain (3):
  - Local Institution, Arganda
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Sweden (4):
  - Local Institution, Halmstad
  - Local Institution, Kungens Kurva
  - Local Institution, Lund
  - Local Institution, Uppsala

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx